CLINICAL TRIAL: NCT02510053
Title: PK-PD of Caspofungin (Cancidas ®) and Drug Tolerance of Fungi to Patients With an Invasive Fungal Infection in the Intensive Care Unit
Brief Title: Pharmacokinetics and Pharmacodynamics of Caspofungin (Cancidas ®) and Drug Tolerance of Fungi to Patients With an Invasive Fungal Infection in the Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhi-jie He, director,clinical research, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14030310568
Record Dates: First submitted 2015-07-19; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Invasive Fungal Infection
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients With IFI in ICU (Other): 40 patients receive Caspofungin for an Invasive Fungal Infection(IFI) in the Intensive Car will be recruited
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — 40 patients with suspected/preoperation/confirmed IFI in ICU received Caspofungin
  Other Names: Cancidas ®

SUMMARY:
To investigate pharmacokinetics(PK) and pharmacodynamics(PD) of Caspofungin in ICU patients after received a loading dose of 70mg followed by 50mg (35mg if Child-Pugh score is 7-9), 40 patients will be recruited. Blood samplings for PK analysis will be collected on day 4 in this study. Caspofungin plasma concentrations are measured by using solid phase extraction and reverse phase high-performance liquid chromatography. Safety analyses will be taken daily during the treatment of Caspofungin. Tests for drug tolerance of fungi and efficacy assessment (clinical and mycological responses) will be taken every 3 days by clinical and mycological tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted to ICU with APACHE-II score more than 15
* Subject is 18 years old and older on the day of the first dosing
* Subject with evidence of proven or probable IFI defined by modified criteria of European Organization for Research and Treatment of Cancer(EORTC)

Exclusion Criteria:

* patient is known to be hypersensitive to caspofungin
* patient's Child-Pugh score is more than 9
* patient is prone to discontinue treatment result from lack of cost
* patient or their guardian refuse to sign a informed consent form
* patient concurrently receiving efavirenz, nevirapine, rifampin, systemic dexamethasone, phenytoin, carbamazepine, phenobarbital, or cyclosporine and other agents have influence on PK parameters of caspofungin
* patient is treated with caspofungin within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | day 4
Area under the plasma concentration versus time curve (AUC) | day 4

SECONDARY OUTCOMES:
Drug-related adverse events | End of caspofungin treatment,an expected average of 20 days